CLINICAL TRIAL: NCT02870062
Title: Impact of Daily Bathing With Chlorhexidine in the Critical Patient: Colonization and Environment
Brief Title: Impact of Daily Bathing With Chlorhexidine in the Critical Patient
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Michel Fernando Martinez-Resendez, M.D., Ph.D., Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IF16-003
Record Dates: First submitted 2016-08-07; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Healthcare Associated Infections
Keywords: Chlorhexidine baths; Critical patient; Healthcare associated infections; Critical care environment; Patient colonization
MeSH Terms: conditions — Cross Infection | interventions — Oral Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine (Experimental): Intervention: daily baths with chlorhexidine wipes, oral spray and shampoo. This arm will receive daily bathing with chlorhexidine wipes at 2% (CLORHEXI-WIPES ONE-STEP, G70 Antisepsis, León, México) plus an oral spray application of chlorhexidine chlorhydrate at 0.12%. For scalp washing, a chlorhexidine shampoo at 0.12% concentration will be applied.
  Interventions: Other: Daily baths with chlorhexidine wipes, oral spray and standard shampoo
- Placebo (Placebo Comparator): Intervention: daily baths with placebo wipes, oral spray and standard shampoo. This arm will receive wipes with the same components as arm #1 plus an oral spray application with the same components except chlorhexidine. For scalp, a standard shampoo will be used. These products will have the same labels and smell as the products in arm #1.
  Interventions: Other: Daily baths with placebo wipes, oral spray and shampoo

INTERVENTIONS:
Other: Daily baths with chlorhexidine wipes, oral spray and standard shampoo — Description already mentioned in arm/group descriptions.
  Other Names: CLORHEXI-WIPES ONE-STEP, G70 Antisepsis
  Arms: Chlorhexidine
Other: Daily baths with placebo wipes, oral spray and shampoo — Description already mentioned in arm/group descriptions.
  Arms: Placebo

SUMMARY:
The search for preventive measure with daily bathing with chlorhexidine in the critical care patient will result in a reduction in patient colonization with multidrug resistant pathogens. Thus, preventing healthcare associated infections. The aim of this study was to determine the impact of daily bathing with chlorhexidine in patient colonization, environment and healthcare workers in the medical intensive care unit (MICU).

The study will be conducted at the University Hospital "Dr. José Eleuterio González", a 450-bed teaching hospital in Monterrey, northeast Mexico.

This is a prospective, experimental, randomized, open-label, double blind study comparing chlorhexidine versus placebo. Any patient 18 years or older admitted to the MICU or with less than 48 hours of patient-days will be included. Patients who present burns with more than 20% body surface, pregnant patients and patients with allergy history to chlorhexidine.

Samples will be obtained from the patient, patient environment and healthcare personnel.

Sampling of the environment (bed rail, mechanical ventilator, table adjacent to the bed, etc.) and patient's anogenital and pharyngeal region will be collected with "swabbing" technique using cotton swabs and cultured according to Public Health England.

Patient skin sampling will be obtained from anorectal region, pharynx, axillary and inguinal fold collected with Williamson-Kligman technique. Colonies will then be further selected and properly cultivated according to their characteristics. Antibiotic susceptibility, clonal relationship, biofilm index and antibiotic susceptibility to chlorhexidine will be determined.

Demographics and clinical data will be collected from admission, throughout hospitalization and discharge.

DETAILED DESCRIPTION:
Introduction:

The search for preventive measure with daily bathing with chlorhexidine in the critical care patient will result in a reduction in patient colonization with multidrug resistant pathogens. Thus, preventing healthcare associated infections. The aim of this study was to determine the impact of daily bathing with chlorhexidine in patient colonization, environment and healthcare workers in the medical intensive care unit (MICU).

Setting:

The study will be conducted at the University Hospital "Dr. José Eleuterio González", a 450-bed teaching hospital in Monterrey, northeast Mexico. The hospital has an average of 22 to 23 thousand yearly discharges with a 20 bed and 15 bed ICU for adults and pediatric/neonatal patients, respectively.

Design and methods:

This is a prospective, experimental, randomized, open-label, double blind study comparing chlorhexidine versus placebo. The randomization will occur 1:1 and the patients will be divided in two groups. The chlorhexidine group will receive daily baths with chlorhexidine wipes at 2% concentration (CLORHEXI-WIPES ONE-STEP, G70 Antisepsis, León, México), plus oral spray with chlorhexidine chlorhydrate at 0.12%. For scalp washing, a chlorhexidine shampoo at 0.12% concentration will be applied. The placebo group, will receive wipes with the same components as arm #1 plus an oral spray application with the same components except chlorhexidine. For scalp, a standard shampoo will be used. These products will have the same labels and smell as the products in the first arm.

Any patient 18 years or older admitted to the MICU or with less than 48 hours of patient-days will be included. Patients who present burns with more than 20% body surface, pregnant patients and patients with allergy history to chlorhexidine. Included patients who develop rash or pruritus after chlorhexidine baths, will be eliminated from the study.

Two weeks previous to the start of the study, MICU personnel will receive theoretical and practical training, were the bathing technique will be taught. Attendance of personnel will be recorded and skills will be surveiled during the intervention.

Bathing technique:

Before use, wipe packages will need to be heated in a conventional microwave for 10-12 seconds, under provider instructions. With the use of globes, the entire skin surface will be covered from the mandibular region to the feet, avoiding contact with mucous membranes such as anal, nasal or urethral membranes. A circular motion will be implemented during bathing.

For facial and genital region, wipes or wet dressings will allowed. The facial and genital region will be the first to clean. Mouthwashes with oral spray solution will be carried out, trying to properly impregnate cheeks, palate, pharynx and tongue, letting the solution sit for a minute before removal.

A towel wipe will be used for the neck and shoulders; using a side of the wipe for the anterior anatomical region and the other side for the posterior region. A wipe will be used for each limb (4 in total), using one side for the anterior region and the back side for the posterior region. A wipe will be designated to the buttocks and perianal region, avoiding the anal region. A wipe will be used for the torso, one for the dorsal region, one for the feet and one will be reserved for spare. For scalp washing, shampoo foam will be applied in a circular motion, trying to cover the entire surface of the scalp, excess will be removed with a dry towels.

Sampling:

Samples will be obtained from the patient and environment. Sampling of the environment (bed rail, mechanical ventilator, table adjacent to the bed, etc.) and patient's anogenital and pharyngeal region will be collected with "swabbing" technique using cotton swabs and cultured according to Public Health England.

Patient skin sampling will be obtained from anorectal region, pharynx, axillary and inguinal fold collected with Williamson-Kligman technique; delimiting an area of 3 cm2 and subsequent application of 1 ml a unionized solution, then proceed to gently scrape the area with a sterile spatula. This liquid is then retrieved with a pipette and cultured directly on a blood agar plate. Colonies will then be further selected and properly cultivated according to their characteristics.

Healthcare personnel samples will also be obtained from pharynx, skin and hands. All these samples will be collected the day of admission to the MICU, first 72 hours, 10th day and once a week until discharge of the patient. In the case of healthcare workers, will be collected at the end of their workday.

Isolate processing:

Samples will be cultured using conventional methods: from prime media, colonies will be taken separately and will be placed in a Brucella broth with 15% glycerol. Specimens will be then frozen to -80ºC.

When processing isolates, conventional phenotypic identification methods will be used. From primary isolate testing, corresponding biochemical tests will be selected for each species identification. When phenotypic tests don't reach isolate identification, molecular based testing and gene amplification will be used.

Antimicrobial susceptibility will be evaluated by the broth microdilution method and according to protocols M07-A10 and M100-S25 from Clinical and Laboratory Standards Institute (CLSI) guidelines and processed by an automatized system (SensititreAris 2X).

Pathogen clonal relationship For clonal relationship, pulsed filed gel electrophoresis will be used. Band pattern will be analyzed visually according to Tenover criteria. Data obtained will be analyzed with statistical software. Polymerase chain reaction (PCR) gene amplification will be obtained to analyze antibiotic resistance patterns for each species.

Pathogen biofilm production:

Biofilm production will be determined by crystal violet staining and a biofilm index will be obtained by spectrophotometry.

Pathogen susceptibility to chlorhexidine:

For determination of minimum inhibitory concentration (MIC) to chlorhexidine, agar dilution method will be applied according to protocol M07-A9 y M100-S20 in CLSI guidelines. Isolates with MIC values of ≥90, will be denoted with reduced susceptibility to such disinfectant.

Clinical data and follow-up:

Demographics and clinical data will be collected from admission, throughout hospitalization and discharge. Variables such as previous hospital admission in the previous year, previous surgeries, history of infection by resistant pathogens, days of hospital stay, instrumentation (use of foley catheter, mechanical ventilation or central venous catheter) and clinical evolution evaluated by Acute Physiology and Chronic Health Evaluation (APACHE-II) and Scale for the Assessment of Positive Symptoms (SAPS).

Positive culture swabs obtained from healthcare workers with resistant pathogens will proceed with reinforcement of hand hygiene and strengthening in universal protection (gloves, face mask, etc). If positive Methicillin-resistant Staphylococcus aureus (MRSA) culture is obtained, intranasal mupirocin treatment will be given for 5 days until a negative culture is achieved.

Hospital Epidemiology team's routine surveillance and monitoring will continue throughout the study period. Rate of healthcare associated infections will be compared to before, during and after intervention. Surveillance of healthcare associated infections will be following Center for Disease Control (CDC) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted to the medical intensive care unit
* Any patient with less than 48 hours in the medical intensive care unit
* Patient's age 18 years or older

Exclusion Criteria:

* Patients with burns greater than 20% body surface
* Pregnancy
* Patients with recorded allergy history to chlorhexidine

Elimination Criteria:

* Patient refuses participation in the study
* Patient develops severe reaction to chlorhexidine, defined as the sudden appearance of rash and/or pruritus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Pathogen colonization | 1 year
  Determine the impact of daily bathing with chlorhexidine in patient colonization, study setting and healthcare workers in the MICU. Patient skin sample and environment swabbing will be collected in day 0 of admission to MICU, day 10 and once a week till discharge. Healthcare worker samples will be collected at the end of every workday. Samples will be cultured using conventional methods: from prime media, colonies will be taken separately and will be placed in a Brucella broth with 15% glycerol and then frozen to -80ºC. When processing isolates, conventional phenotypic identification methods will be used.
  Antimicrobial susceptibility will be evaluated by the broth microdilution method according to CLSI guidelines and processed by an automatized system (SensititreAris 2X).

SECONDARY OUTCOMES:
Healthcare associated infections | 1 year
  Determine if chlorhexidine baths have an effect on healthcare associated infections. Hospital Epidemiology team's routine surveillance and monitoring will continue throughout the study period. Rate of healthcare associated infections will be compared to before, during and after intervention.
Pathogen clonal relationship | 1 year
  After specimen identification using conventional methods, pathogen clonal relationship will be obtained. For clonal relationship, pulsed filed gel electrophoresis will be used. Band pattern will be analyzed visually according to Tenover criteria. Data obtained will be analyzed with statistical software. PCR gene amplification will be obtained to analyze antibiotic resistance patterns for each species.
Pathogen biofilm index | 1 year
  After specimen identification using conventional methods, pathogen biofilm index will also be obtained. Biofilm production will be determined by crystal violet staining and a biofilm index will be obtained by spectrophotometry.
Pathogen susceptibility to chlorhexidine | 1 year
  For determination of minimum inhibitory concentration (MIC) to chlorhexidine, agar dilution method will be applied according to protocol M07-A9 y M100-S20 in CLSI guidelines. Isolates with MIC values of ≥90, will be denoted with reduced susceptibility to such disinfectant.

CONTACTS AND LOCATIONS:
Overall Officials: Michel F Martinez-Resendez, M.D., Principal Investigator — Associate Professor of Infectious Diseases

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available. Individual data will remain confidential, according to our ethical committee regulations.

REFERENCES:
- [Background] Williamson P, Kligman AM. A new method for the quantitative investigation of cutaneous bacteria. J Invest Dermatol. 1965 Dec;45(6):498-503. doi: 10.1038/jid.1965.164. No abstract available. PMID 5321315
- [Background] Tenover FC, Arbeit RD, Goering RV, Mickelsen PA, Murray BE, Persing DH, Swaminathan B. Interpreting chromosomal DNA restriction patterns produced by pulsed-field gel electrophoresis: criteria for bacterial strain typing. J Clin Microbiol. 1995 Sep;33(9):2233-9. doi: 10.1128/jcm.33.9.2233-2239.1995. No abstract available. PMID 7494007
- [Background] Christensen GD, Simpson WA, Younger JJ, Baddour LM, Barrett FF, Melton DM, Beachey EH. Adherence of coagulase-negative staphylococci to plastic tissue culture plates: a quantitative model for the adherence of staphylococci to medical devices. J Clin Microbiol. 1985 Dec;22(6):996-1006. doi: 10.1128/jcm.22.6.996-1006.1985. PMID 3905855